CLINICAL TRIAL: NCT04660032
Title: Randomized Evaluation of Hypertensive Moms: Interventional Nudge to Drive Transitions of Care
Brief Title: Nudge to Drive Transitions of Care
Acronym: REMIND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 844269
Record Dates: First submitted 2020-12-02; First posted 2020-12-09 (Actual); Results first posted 2024-08-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-02

CONDITIONS: Preeclampsia; Preeclampsia Severe; Gestational Hypertension; Hypertensive Disorder of Pregnancy; Superimposed Pre-Eclampsia
Keywords: Nudge; Postpartum; Fourth trimester; Cardiovascular disease
MeSH Terms: conditions — Pre-Eclampsia; Hypertension, Pregnancy-Induced; Toxemia; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant
Masking Description: The participant will be unaware of whether their obstetric provider received an electronic prompt.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nudge (Experimental): Obstetric care providers will receive electronic prompts (nudge) for participants in this arm
  Interventions: Behavioral: Nudge
- Usual care (No Intervention): Usual postpartum follow-up with visit at 4-12 weeks postpartum

INTERVENTIONS:
Behavioral: Nudge — An electronic prompt (nudge) will be sent to the participant's obstetric care provider. The provider will receive a staff message in Epic (Penn Chart) that his/her patient has an upcoming postpartum visit. The message will be sent 1 week before the scheduled visit. The message will have patient-specific information including hypertensive diagnosis, blood pressure medication(s), gestational diabetes diagnosis, and primary care provider as listed in the Epic banner. The message will also have dot phrases for recommended counseling and contact information for UPHS primary care and cardiology providers. There will be example text recommending follow-up with primary care or cardiology; counseling on risk of future CVD; and recommending aspirin in a future pregnancy.
  Arms: Nudge

SUMMARY:
Hypertensive disorders of pregnancy (HDP) are stress tests which may identify women at high risk of future cardiovascular disease (CVD), the leading cause of death among women. Given the public health impact of HDP and CVD, there is a compelling need to identify scalable interventions to improve preventative care among women who have risk identified during pregnancy. We will examine the effects of delivering electronic prompts to obstetric care providers (nudge) on transitions of care in the postpartum period. We will conduct a pilot randomized trial to evaluate whether this nudge intervention will improve postpartum counseling and lead to greater follow-up with preventative care providers among women with HDP.

DETAILED DESCRIPTION:
Background:

Women with HDP need ongoing care in the postpartum and inter-pregnancy period. HDP, including preeclampsia (PEC) and gestational hypertension (GHTN), complicate up to 10% of all pregnancies and are associated with immediate and long-term cardiovascular morbidity and mortality. HDP increase lifelong risk for chronic hypertension, diabetes, ischemic heart disease, stroke, and heart failure. Black women have a higher incidence of HDP and have a disproportionately higher morbidity and mortality compared to non-black women. The American College of Obstetricians and Gynecologists (ACOG) and the American Heart Association (AHA) emphasize the postpartum period as an important opportunity to identify and intervene upon women at high-risk for future cardiovascular disease (CVD).

However, current postpartum practices inadequately address transitions of care for women with HDP. A significant proportion of women with HDP do not see a preventative care provider (primary care, cardiology) in the months after delivery. Black women are particularly vulnerable to being lost to follow-up after complicated pregnancy. The HSM program is an innovative, patient-centered program that monitors postpartum blood pressure remotely using a text-based interface. It is supported by the Way to Health platform. HSM improves blood pressure management in the two weeks after delivery and eliminates racial disparities in blood pressure ascertainment during that time. However, enrollment in HSM did not improve follow-up in the year after delivery, with less than 1/3 of women having a preventative care visit. Poor follow-up is likely multifactorial, but may be driven by inadequate patient counseling in the postpartum period. Among women enrolled in HSM, only 21% of women were counseled on follow-up with primary care and only 4% were counseled on CVD risk at their postpartum visits based on chart review.

Nudges are effective for changing medical decision-making and improving clinical outcomes. Nudges utilize concepts from behavioral economics to subtly change the decision-making environment to facilitate evidence-based care and can be delivered to patients, providers, or both. Examples of nudges include electronic prompts to order cancer screening and electronic defaults that guide ordering practices. Nudges are low cost, scalable using Electronic Medical Record (EMR) systems, and improve rates of preventative services including influenza vaccination, referral to mammography, and statin prescription for CVD prevention.

Design:

This study will use a randomized, controlled superiority trial to evaluate a hospital-wide initiative to improve counseling for postpartum women who experienced HDP during their pregnancy or in the immediate postpartum period.

Hypotheses:

1. The investigators hypothesize that the prompt will increase the proportion of women counseled on transitioning care to a primary care provider or cardiologist after pregnancy (primary outcome).
2. The investigators hypothesize that the provider nudge will increase the proportion of women attending a preventative care visit within 6 months of delivery as assessed by chart review and patient surveys.

The HSM daily log generated through the Way to Health platform will be used to generate lists of patients who are eligible for the study. For each eligible woman, the date of and obstetric care provider for her postpartum visit will be recorded within 3 weeks of delivery.

Patients will then be randomly assigned to a control group with no intervention (usual care through HSM) or the intervention group (physician nudge) using simple 1:1 randomization through the Way to Health Platform. If a woman is randomized to the intervention arm, her obstetric care provider for her postpartum visit will receive a staff message in Epic (Penn Chart) that the provider's patient has an upcoming postpartum visit. The message will be sent 1 week before the scheduled visit. The message will have patient-specific information including hypertensive diagnosis, blood pressure medication(s), gestational diabetes diagnosis, and primary care provider as listed in the Epic banner. The message will also have dot phrases for recommended counseling and contact information for University of Pennsylvania Health System (UPHS) primary care and cardiology providers. There will be a dot phrase recommending follow-up with primary care or cardiology; counseling on risk of future CVD; and recommending aspirin in a future pregnancy.

A web-based survey will be distributed to all women in the study 6 months after delivery through the Way to Health platform. The survey will assess attendance at a preventative care visit, social determinants of health, health status, and insurance status after delivery.

Demographic characteristics, medical and obstetric history, hypertensive disorder, laboratory test results (platelet count, creatinine, liver function tests, urine protein, total cholesterol, triglycerides, LDL-C, HDL-C, glucose, hemoglobin A1c), blood pressure measurements, height, weight, and office visits within 6 months of delivery will be abstracted from the EMR. Detailed chart abstraction will be performed regarding counseling at the postpartum visit and additional office visits within 6 months of delivery focusing on 1) health maintenance 2) hypertension, or 3) cardiovascular risk reduction. Two reviewers will assess counseling at each visit. The investigators will obtain data on obstetric care providers including level (resident physician, attending physician, nurse practitioner, physician assistant, or certified nurse midwife), gender, and years in practice from publicly available databases or websites online.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years old.
2. Have a diagnosis of HDP during delivery admission or have a diagnosis made at time of evaluation in the Perinatal Evaluation and Treatment Unit after discharge from the delivery admission. HDP diagnoses are based on criteria from the American College of Obstetricians and Gynecologists (ACOG).
3. Enrolled in Heart Safe Motherhood at Pennsylvania Hospital.
4. Have a postpartum visit with a University of Pennsylvania HealthSystem provider scheduled 4-12 weeks after delivery.

Exclusion Criteria:

1. Women diagnosed with chronic hypertension (CHTN) without superimposed pre-eclampsia (PEC).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2022-06-22 (Actual); Study Completion 2023-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jourdan E Triebwasser, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Pennsylvania Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hutcheon JA, Lisonkova S, Joseph KS. Epidemiology of pre-eclampsia and the other hypertensive disorders of pregnancy. Best Pract Res Clin Obstet Gynaecol. 2011 Aug;25(4):391-403. doi: 10.1016/j.bpobgyn.2011.01.006. Epub 2011 Feb 18. PMID 21333604
- [Background] Timpka S, Stuart JJ, Tanz LJ, Rimm EB, Franks PW, Rich-Edwards JW. Lifestyle in progression from hypertensive disorders of pregnancy to chronic hypertension in Nurses' Health Study II: observational cohort study. BMJ. 2017 Jul 12;358:j3024. doi: 10.1136/bmj.j3024. PMID 28701338
- [Background] Cirillo PM, Cohn BA. Pregnancy complications and cardiovascular disease death: 50-year follow-up of the Child Health and Development Studies pregnancy cohort. Circulation. 2015 Sep 29;132(13):1234-42. doi: 10.1161/CIRCULATIONAHA.113.003901. Epub 2015 Sep 21. PMID 26391409
- [Background] Theilen LH, Fraser A, Hollingshaus MS, Schliep KC, Varner MW, Smith KR, Esplin MS. All-Cause and Cause-Specific Mortality After Hypertensive Disease of Pregnancy. Obstet Gynecol. 2016 Aug;128(2):238-244. doi: 10.1097/AOG.0000000000001534. PMID 27400006
- [Background] Wu P, Haththotuwa R, Kwok CS, Babu A, Kotronias RA, Rushton C, Zaman A, Fryer AA, Kadam U, Chew-Graham CA, Mamas MA. Preeclampsia and Future Cardiovascular Health: A Systematic Review and Meta-Analysis. Circ Cardiovasc Qual Outcomes. 2017 Feb;10(2):e003497. doi: 10.1161/CIRCOUTCOMES.116.003497. Epub 2017 Feb 22. PMID 28228456
- [Background] Gyamfi-Bannerman C, Pandita A, Miller EC, Boehme AK, Wright JD, Siddiq Z, D'Alton ME, Friedman AM. Preeclampsia outcomes at delivery and race. J Matern Fetal Neonatal Med. 2020 Nov;33(21):3619-3626. doi: 10.1080/14767058.2019.1581522. Epub 2019 Feb 20. PMID 30786794
- [Background] Miranda ML, Swamy GK, Edwards S, Maxson P, Gelfand A, James S. Disparities in maternal hypertension and pregnancy outcomes: evidence from North Carolina, 1994-2003. Public Health Rep. 2010 Jul-Aug;125(4):579-87. doi: 10.1177/003335491012500413. PMID 20597458
- [Background] ACOG Committee Opinion No. 736: Optimizing Postpartum Care. Obstet Gynecol. 2018 May;131(5):e140-e150. doi: 10.1097/AOG.0000000000002633. PMID 29683911
- [Background] Brown HL, Warner JJ, Gianos E, Gulati M, Hill AJ, Hollier LM, Rosen SE, Rosser ML, Wenger NK; American Heart Association and the American College of Obstetricians and Gynecologists. Promoting Risk Identification and Reduction of Cardiovascular Disease in Women Through Collaboration With Obstetricians and Gynecologists: A Presidential Advisory From the American Heart Association and the American College of Obstetricians and Gynecologists. Circulation. 2018 Jun 12;137(24):e843-e852. doi: 10.1161/CIR.0000000000000582. Epub 2018 May 10. No abstract available. PMID 29748185
- [Background] Bennett WL, Chang HY, Levine DM, Wang L, Neale D, Werner EF, Clark JM. Utilization of primary and obstetric care after medically complicated pregnancies: an analysis of medical claims data. J Gen Intern Med. 2014 Apr;29(4):636-45. doi: 10.1007/s11606-013-2744-2. Epub 2014 Jan 29. PMID 24474651
- [Background] Levine LD, Nkonde-Price C, Limaye M, Srinivas SK. Factors associated with postpartum follow-up and persistent hypertension among women with severe preeclampsia. J Perinatol. 2016 Dec;36(12):1079-1082. doi: 10.1038/jp.2016.137. Epub 2016 Sep 1. PMID 27583396
- [Background] Lewey J, Levine LD, Yang L, Triebwasser JE, Groeneveld PW. Patterns of Postpartum Ambulatory Care Follow-up Care Among Women With Hypertensive Disorders of Pregnancy. J Am Heart Assoc. 2020 Sep;9(17):e016357. doi: 10.1161/JAHA.120.016357. Epub 2020 Aug 27. PMID 32851901
- [Background] Hirshberg A, Downes K, Srinivas S. Comparing standard office-based follow-up with text-based remote monitoring in the management of postpartum hypertension: a randomised clinical trial. BMJ Qual Saf. 2018 Nov;27(11):871-877. doi: 10.1136/bmjqs-2018-007837. Epub 2018 Apr 27. PMID 29703800
- [Background] Hirshberg A, Sammel MD, Srinivas SK. Text message remote monitoring reduced racial disparities in postpartum blood pressure ascertainment. Am J Obstet Gynecol. 2019 Sep;221(3):283-285. doi: 10.1016/j.ajog.2019.05.011. Epub 2019 May 20. No abstract available. PMID 31121137
- [Background] Patel MS. Nudges for influenza vaccination. Nat Hum Behav. 2018 Oct;2(10):720-721. doi: 10.1038/s41562-018-0445-x. No abstract available. PMID 31406293
- [Background] Patel MS, Navathe AS, Liao JM. Using Nudges to Improve Value by Increasing Imaging-Based Cancer Screening. J Am Coll Radiol. 2020 Jan;17(1 Pt A):38-41. doi: 10.1016/j.jacr.2019.08.025. Epub 2019 Sep 18. No abstract available. PMID 31541658
- [Background] Patel MS, Volpp KG, Small DS, Wynne C, Zhu J, Yang L, Honeywell S Jr, Day SC. Using Active Choice Within the Electronic Health Record to Increase Influenza Vaccination Rates. J Gen Intern Med. 2017 Jul;32(7):790-795. doi: 10.1007/s11606-017-4046-6. Epub 2017 Mar 23. PMID 28337690
- [Background] Yokum D, Lauffenburger JC, Ghazinouri R, Choudhry NK. Letters designed with behavioural science increase influenza vaccination in Medicare beneficiaries. Nat Hum Behav. 2018 Oct;2(10):743-749. doi: 10.1038/s41562-018-0432-2. Epub 2018 Oct 1. PMID 31406294
- [Background] Hsiang EY, Mehta SJ, Small DS, Rareshide CAL, Snider CK, Day SC, Patel MS. Association of an Active Choice Intervention in the Electronic Health Record Directed to Medical Assistants With Clinician Ordering and Patient Completion of Breast and Colorectal Cancer Screening Tests. JAMA Netw Open. 2019 Nov 1;2(11):e1915619. doi: 10.1001/jamanetworkopen.2019.15619. PMID 31730186
- [Background] Patel MS, Kurtzman GW, Kannan S, Small DS, Morris A, Honeywell S Jr, Leri D, Rareshide CAL, Day SC, Mahoney KB, Volpp KG, Asch DA. Effect of an Automated Patient Dashboard Using Active Choice and Peer Comparison Performance Feedback to Physicians on Statin Prescribing: The PRESCRIBE Cluster Randomized Clinical Trial. JAMA Netw Open. 2018 Jul 6;1(3):e180818. doi: 10.1001/jamanetworkopen.2018.0818. PMID 30646039
- [Derived] Triebwasser JE, Lewey J, Walheim L, Sehdev HM, Srinivas SK. Electronic Reminder to Transition Care After Hypertensive Disorders of Pregnancy: A Randomized Controlled Trial. Obstet Gynecol. 2023 Jul 1;142(1):91-98. doi: 10.1097/AOG.0000000000005237. Epub 2023 Jun 7. PMID 37294089

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nudge | Usual Care
Started | 105 | 119
Completed | 104 | 118
Not Completed | 1 | 1
Not completed — Protocol Violation | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nudge | Usual Care | Total
Number analyzed (Participants) | 104 | 118 | 222
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.0 (5.5) | 32.7 (5.2) | 32.3 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104 | 118 | 222
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 4 | 7 | 11
  Black | 34 | 31 | 65
  Hispanic or Latinx | 7 | 6 | 13
  Multiple races/ethnicities | 2 | 4 | 6
  Not Reported | 0 | 3 | 3
  White | 57 | 67 | 124
Region of Enrollment [Number; unit: participants]
  United States | 104 | 118 | 222
Public insurance [Count of Participants; unit: Participants] | 32 | 37 | 69
Body mass index at first prenatal visit [Median (Inter-Quartile Range); unit: kg/m^2] | 28.0 [23.8 to 33.2] | 27.5 [23.9 to 32.7] | 27.8 [23.9 to 33.1]
Nulliparity [Count of Participants; unit: Participants] | 64 | 69 | 133
History of hypertensive disorder of pregnancy [Count of Participants; unit: Participants] | 22 | 32 | 54
Chronic hypertension [Count of Participants; unit: Participants] | 9 | 14 | 23
Diabetes [Count of Participants; unit: Participants] — Pregestational or gestational diabetes
  Participants | 7 | 19 | 26
Tobacco use [Count of Participants; unit: Participants] | 5 | 5 | 10
Gestational age at delivery (weeks) [Median (Inter-Quartile Range); unit: weeks] | 38.5 [37.4 to 39.9] | 38.5 [37.4 to 39.6] | 38.5 [37.4 to 39.7]
Hypertensive disorder of pregnancy [Count of Participants; unit: Participants]
  Gestational hypertension or preeclampsia | 75 | 85 | 160
  Preeclampsia with severe features | 20 | 19 | 39
  Hemolysis, elevated liver enzymes, and low platelet (HELLP) syndrome | 0 | 1 | 1
  Chronic hypertension with superimposed preeclampsia | 9 | 13 | 22

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Documented Counseling on Transitions of Care
Description: The primary outcome measure is documentation of counseling about transitioning care to a continuity care provider (primary care or cardiology) at the postpartum visit.
Time Frame: 4-12 weeks postpartum
Population: Analyzed for study participants who attended postpartum visit
Measure: Count of Participants; unit: Participants
Arm/Group | Nudge | Usual Care
Number analyzed (Participants) | 98 | 107
Participants | 38 | 28

2. Secondary Outcome: Nudge Message Opened Within 1 Week of Receipt
Description: Electronic prompts opened by obstetric care providers within 1 week of receipt in the electronic medical record. The nudge (electronic prompt) was sent 1 week prior to the scheduled 4-12 weeks postpartum visit.
Time Frame: Prior to postpartum visit
Population: A nudge was only sent for the intervention group; it was not sent nor measured for usual care.
  A single nudge message was sent to the scheduled postpartum care provider per patient in the intervention group. A single provider could receive more than 1 nudge if they had more than 1 patient who was included in the study.
Measure: Count of Units; unit: Nudge
Units Other Than Participants: Nudge
Arm/Group | Nudge | Usual Care
Number analyzed (Participants) | 104 | 0
Number analyzed (Nudge) | 104 | 0
Nudge | 104 | 0

3. Secondary Outcome: Number of Patients With Documented Counseling on Cardiovascular Disease (CVD) Risk at the Postpartum Visit
Description: Documentation in the postpartum visit note regarding ongoing cardiovascular risk related to HDP
Time Frame: 4-12 weeks postpartum
Population: 98 of 104 patients in the nudge arm (6 lost to follow-up) and 107 of 118 (11 lost to follow-up) patients in the usual care arm attended a postpartum visit within the health system and could be evaluated for this secondary outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Nudge | Usual Care
Number analyzed (Participants) | 98 | 107
Participants | 21 | 9

4. Secondary Outcome: Number of Participants With Postpartum Visit Notes That Used Example Text
Description: Use of scripted dot phrases (available in Epic) for counseling on transitions of care and CVD risk in the postpartum note. These dot phrases were available for all providers and were included in the nudge message.
Time Frame: 4-12 weeks postpartum
Population: Attended postpartum visit
Measure: Count of Participants; unit: Participants
Arm/Group | Nudge | Usual Care
Number analyzed (Participants) | 98 | 107
Participants | 11 | 1

5. Secondary Outcome: Number of Patients With Preventative Care Follow-up
Description: Attendance at a primary care or cardiology visit for preventative care within 6 months of delivery.
Time Frame: 6 months postpartum
Population: Entire enrolled population who met inclusion/exclusion criteria
Measure: Count of Participants; unit: Participants
Arm/Group | Nudge | Usual Care
Number analyzed (Participants) | 104 | 118
Participants | 23 | 29

ADVERSE EVENTS:
Time Frame: Adverse events were not assessed as the intervention was a message to providers and not a direct intervention with patients.
Description: Adverse events were not assessed as the intervention was a message to providers and not a direct intervention with patients.
Arm/Group | Nudge | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-21): https://cdn.clinicaltrials.gov/large-docs/32/NCT04660032/Prot_SAP_000.pdf